CLINICAL TRIAL: NCT07342998
Title: Could Computerized Tomography (CT) Scans be Used as an Alternative to Colonoscopies for Colorectal Cancer Screenings?
Brief Title: Could Computerized Tomography be an Alternative to Colonoscopies for Screening for Colorectal Cancer?
Status: Active, not recruiting | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Mucahit UNAL, Assistant Professor, Bilecik Seyh Edebali Universitesi
Other Study IDs: E-10333602-050.04-339197
Record Dates: First submitted 2025-12-21; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Colo-rectal Cancer; Screening Colonscopy; Colon Cancer Screening
Keywords: colonscopy; colon cancer; cancer screening
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- colonscopy: participant screened by colonoscopy
- tomography: participant screened by tomography

SUMMARY:
The aim of this observational study is to investigate whether computed tomography can be used as an alternative to colonoscopy in colon cancer screening. The main question the study aims to answer is:

Can colon cancer screening be performed as effectively with computed tomography as with colonoscopy?

Participants in the colon cancer screening group will be divided into two groups: those who underwent colonoscopy and those who underwent computed tomography. The screening effectiveness of the two methods will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All participants aged 50-70 who have undergone colonoscopy screening
* All participants aged 50-70 who have undergone abdominal computed tomography

Exclusion Criteria:

- The patient has a history of colon cancer

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CT scans and colonoscopies performed on patients aged 50-70 at Bilecik Research and Training Hospital between January 1, 2023, and December 31, 2024, will be examined.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
polyp/cancer incidance | when the pathology results are available after a colonoscopy or when the report is written after a CT scan through study completion, an average of 2 years
  Number of patients with polyps and cancer detected by screening

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Seyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mang T, Graser A, Schima W, Maier A. CT colonography: techniques, indications, findings. Eur J Radiol. 2007 Mar;61(3):388-99. doi: 10.1016/j.ejrad.2006.11.019. Epub 2007 Jan 16. PMID 17224254
- [Result] Iwatsuki K, Murakami T, Manabe Y, Narai H, Warita H, Hayashi T, Abe K. Two cases of Japanese CADASIL with corpus callosum lesion. Tohoku J Exp Med. 2001 Oct;195(2):135-40. doi: 10.1620/tjem.195.135. PMID 11846209